CLINICAL TRIAL: NCT05446597
Title: Symptom Management vs Alternative Randomized Treatment of Concussion Trial
Brief Title: SMART Concussion Trial: Symptom Management vs Alternative Randomized Treatment of Concussion Trial
Acronym: SMART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB21-1045
Record Dates: First submitted 2022-06-07; First posted 2022-07-06 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Mild Traumatic Brain Injury; Headaches Posttraumatic; Neck Pain; Dizziness
MeSH Terms: conditions — Brain Concussion; Post-Traumatic Headache; Neck Pain; Dizziness

STUDY DESIGN:
Intervention Model Description: This is a single-blind randomized controlled superiority trial with three treatment groups. Trial participants will be screened for headache and neck pain/dizziness based on symptom ratings on the Sport Concussion Assessment Tool 5 (SCAT5) Post-Concussion Symptom Scale (PCSS) (rating 0-2 mild, 3-4 moderate, 5-6 severe /6). Patients will be allocated to one of three treatments based on symptom severity:
  1. Headache treatment
  2. Neck pain / Dizziness treatment
  3. Multimodal treatment All participants will receive standard of care education and exercise recommendations based on BCTT and sub-symptom threshold tolerance at baseline
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Headache Treatment (Experimental): Participants in the headache arm will be randomized to receive a peripheral, greater occipital nerve block with 0.5% Bupivacaine or the multimodal treatment protocol. Participants will complete a daily headache diary over the 6-week treatment period, following a link on their mobile device. Patients receiving a nerve block will have weekly over-the-phone or virtual check-ins by the study team to evaluate for any side effects, pain, as needed medications, and study compliance. These patients will be given supplemental HA education as needed. Participants receiving the block will be offered a second block at 6 weeks if they meet the following criteria: a. no side effects with the first block, b. participant received relief from the first block and prefers a second, and c. headache is still occurring at least once per week. Participants randomized to the multimodal treatment portion, will have up to 6 weeks of scheduled multimodal treatment sessions.
  Interventions: Procedure: Symptom-specific Headache Treatment; Behavioral: Multimodal Concussion Treatment
- Dizziness and/or Neck Pain Treatment (Experimental): Participants will be randomized to receive cervicovestibular physiotherapy (CV PT) or the multimodal treatment program. The CV PT group will participate in a combination of cervical spine and vestibular rehabilitation as per a standardized treatment algorithm based on individual assessment findings for six weeks. This form of therapy combines treatment techniques for both the cervical spine and vestibular system that are commonly used in physiotherapy practice. Cervical spine treatments may include neuromotor retraining, sensorimotor retraining, manual therapy, soft tissue techniques, and range of motion exercises. Vestibular rehabilitation may include gaze stabilization, habituation, standing balance, and dynamic balance.
  Interventions: Other: Symptom-specific Dizziness &/or Neck Pain Treatment; Behavioral: Multimodal Concussion Treatment
- Multimodal Treatment (Experimental): The multimodal treatment consists of 6 treatment sessions that will combine basic physiotherapy exercises to address dizziness and balance problems, training in deep breathing, progressive muscle relaxation, visualization to address headache, sleep hygiene education to address insomnia, and cognitive-behavioral intervention and gratitude exercises to promote coping and resilience. The treatment is designed to be implemented by a variety of clinical health care professionals.
  Interventions: Behavioral: Multimodal Concussion Treatment

INTERVENTIONS:
Procedure: Symptom-specific Headache Treatment — Greater Occipital Nerve Block
  Arms: Headache Treatment
Other: Symptom-specific Dizziness &/or Neck Pain Treatment — Cervicovestibular Physiotherapy Treatment
  Arms: Dizziness and/or Neck Pain Treatment
Behavioral: Multimodal Concussion Treatment — Lite combination of headache advice, general physiotherapy exercises, mindfulness, visualization, and relaxation

SUMMARY:
Given the rising rates of concussion in youth ages 10-19 and the significant proportion of young people who remain symptomatic for months following concussion, research evaluating the efficacy of multifaceted treatment options following concussion is imperative. Studies examining the efficacy of treatment strategies following concussion in children and adults are surprisingly limited, and most focus on one treatment approach, have small sample sizes, are not randomized controlled trials, and focus on individuals with prolonged recovery (months). There is a need for a multifaceted treatment trial to examine the early implementation of treatment approaches that may reduce prolonged recovery while considering the heterogeneous presentation of symptoms and patient preferences in the sub-acute stage following concussion. Randomized controlled trials that consider a multifaceted transdisciplinary approach to treatment in the early period following concussion are needed to raise the bar regarding evidence-informed management following concussion

DETAILED DESCRIPTION:
The primary objective of this RCT is to examine if up to 6-weeks of symptom-specific (1. headache, 2. dizziness and/or neck pain) treatment initiated in the acute/sub-acute stages following concussion in 13-19 year-old participants recruited acutely (within 2 weeks) following concussion are superior to up to 6 weeks of a multimodal, non-symptom specific treatment program. Treatment will cease once participants are cleared to return to unrestricted physical activity by a sports medicine physician, and will therefore last up to 6 weeks. We have two primary outcomes:

1. Post-Concussion Total Symptom Score (PCSS /132) on the SCAT5 following treatment of up to six sessions
2. Days from injury to physician clearance to return to unrestricted physical activity (e.g., physical education, sport, recreational activities)

ELIGIBILITY:
Inclusion Criteria:

* 13 - 19 years of age at the start of treatment
* Diagnosed by the study physician with a concussion as per the 5th International Consensus Statement on Concussion in Sport1
* Glasgow Coma Scale 13-15 if recorded
* Loss of consciousness < 30 minutes if present
* Post-traumatic amnesia < 24 hours if present
* Diagnosis within 2 weeks of injury
* Moderate-severe symptoms of dizziness, neck pain, headaches, or sleep disturbance at > one week and < three weeks post injury reported on the PCSS (3-6 on 0-6 Likert scale for at least one of three symptoms)
* Patients can have a history of migraine or a family history of migraine

Exclusion Criteria:

* Inability to communicate orally and/or in writing in English language
* Significant developmental delay or intellectual disability
* No access to smartphone or computer
* Red flags or other clinical indication suggesting that further medical investigation is warranted (e.g., neurological scan - reflexes, dermatomes, myotomes, long tract signs, CN II-XII, Cerebellar Scan
* Unresolved Benign Paroxysmal Positional Vertigo (BPPV) (Dix-Hallpike and Roll Test)
* Inability to participate in physical activity for a reason other than concussion
* Orthopedic or other injury precluding ability to participate
* Medical history of neurological conditions: seizures (febrile SZ will be allowed), stroke, previous moderate/severe TBI, CNS cancers, SCI
* Psychotic disorder
* Inability to provide informed consent
* History of surgery in the occipital region
* Uncontrolled rheumatologic, inflammatory, or neurologic disorders (eg MS); Fibromyalgia/chronic fatigue syndrome; coagulopathy; immunosuppression
* Active cancer
* Herpes zoster infection in last 6 months
* Pregnancy
* Steroid injection to the greater or lesser occipital nerve infiltration in past 3 months
* Previously enrolled in the trial

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms | Collected at 6 weeks from the start of treatment
  Change from baseline in symptom burden, measured by the Post-Concussion Symptom Score (PCSS /132) on the SCAT5 (Sport Concussion Assessment Tool - 5th Edition) at 6 weeks following initiation of treatment. Options for scores are: none (0), mild (1), moderate (2), or severe (3) in 22 symptom categories, for a total score of 0 (no symptoms) to 132 (severe symptoms in all categories)
Return to unrestricted physical activity | Measured until 3 months from the start of treatment
  Days from injury to physician clearance to return to unrestricted physical activity (e.g., physical education, sport, recreational activities)

SECONDARY OUTCOMES:
Change in symptoms on the Buffalo Concussion Treadmill Test | Measured at 6 weeks from the start of treatment
  Change in overall symptoms [visual analogue scale (VAS) 0-10] from rest prior to the Buffalo Concussion Treadmill Test (BCTT) to age-predicted 80% maximum heart rate on the BCTT at 6-weeks. 0 indicates 'Feeling Good' up to 10 'Worst I have ever felt'.
Changes in symptom-specific ratings | Measured at 6 weeks from the start of treatment
  Symptom-specific PCSS [Post-Concussion Symptom Score (PCSS /132)] ratings of headache, dizziness/neck pain, and sleep disturbance [0-6 Likert scale; from no symptoms (0), to moderate (3), to severe (6)]
Change in quality of life rating | Measured at 6 weeks from the start of treatment
  Pediatric Quality of Life Inventory V4.0 (PedsQL) at 6-weeks. Likert scale: never a problem (0) to sometimes (2) to almost always (4). Total symptom scores from 0/94 up to 94/94. Higher scores indicate poorer quality of life
Change in resilience | Measured at 6 weeks from the start of treatment
  Resilience at 6-weeks using the short, 10-item Connor-Davidson Resilience Scale (CD-RISC). Respondents rate items on a 5-point Likert scale, ranging from 0 (not true at all) to 4 (true nearly all the time) for a score range of 0-40. A higher score indicates higher resilience

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Emery, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT05446597/ICF_000.pdf